CLINICAL TRIAL: NCT05585008
Title: Three Dimensional Printed Versus Conventional Heat Cured Acrylic Complete Denture: An In-Vivo Comparative Study
Brief Title: Three Dimensional Printed Versus Conventional Heat Cured Acrylic Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 318/2021
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Completely Edentulous Patients
Keywords: 3d printing; CAD-CAM; retention; adaptation; denture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): group A will receive a conventional heat-cure acrylic denture
  Interventions: Device: two different denture manufacturing technique (heat cure pack and press technique(heat cure acrylic,Acrostone,Egypt)/3d printed dneture(HARZ lab,Russia))
- group B (Active Comparator): group B will receive a 3D printed complete denture
  Interventions: Device: two different denture manufacturing technique (heat cure pack and press technique(heat cure acrylic,Acrostone,Egypt)/3d printed dneture(HARZ lab,Russia))

INTERVENTIONS:
Device: two different denture manufacturing technique (heat cure pack and press technique(heat cure acrylic,Acrostone,Egypt)/3d printed dneture(HARZ lab,Russia)) — retention for the two groups will be measured at 0,1 and 3months, patient satisfaction will be recorded, and accuracy of the denture base will be measured on the software.

SUMMARY:
Introduction:

One major complaint frequently voiced by complete denture wearers is denture retention. Conventional denture disadvantage is heat-curing resin deformation. In addition, the pack and press technique that is still more common, residual stresses that occur at the time of packing are released when the material is removed from the flask, causing the resin to shrink, and this shrinkage is cited as a cause of poor fit of the denture base, In the field of prosthetic dentistry, the ability of additive manufacturing to fabricate prosthetic devices based on CAD data influences the overall quality, the mechanical properties of printed parts, the total cost and the manufacturing time. The milling process wastes large quantities of denture base material, and more recent three-dimensional (3D) prototyping promises a more sustainable additive approach by using less denture resin. However, no clinical reports have been published regarding the accuracy of the mucosal surface or denture retention for denture fabricated using conventional techniques compared to those fabricated using additive manufacturing.

Aim of the study:

Investigate the effect of two techniques of complete denture manufacturing (conventional and 3D printed) on denture retention, trueness (accuracy), and satisfaction.

Methodology:

Twenty patients will be selected from the outpatient clinic and will be divided into 2 groups, group A for conventional dentures and group B for 3D printed dentures, retention for the two groups will be measured at 0,1 and 3 months, and patient satisfaction will be recorded, and accuracy of the denture base will be measured on the software. The results will be tabulated and statistically analyzed using the SPSS program.

DETAILED DESCRIPTION:
Twenty patients will be selected from the Faculty of Dentistry (Suez Canal University) outpatient clinics with the following criteria:

* Patients with good neuromuscular control and free of systemic diseases
* Well-formed ridges with firm and healthy mucosa and no bilateral anterior undercuts.

The patients will be divided equally into two groups(n=10), group (A) which will receive conventional heat cure acrylic denture, and group (B) which will receive 3D printed denture.

Methodology:

A primary impression will be taken for each patient and a special self-cured acrylic tray will be fabricated.

Zinc oxide secondary impression (caves outline, Cavex Holland)will be taken for each patient. The impression will be poured with extra hard stone and labeled master cast.

The cast will be scanned and saved in standard tessellation language (stl) format (master cats).

Jaw relation records for each patient will be taken in the conventional method. For group A: the setting up of teeth will be done in a conventional way on the articulator, and flasking of the waxed-up denture will be done. Wax elimination will be done then packing of heat cure acrylic will be done.

For group B: occlusion block will be scanned (swing scanner, DOF inc, Korea)(the scanner has an accuracy of 10 μm) after taking jaw relation record.

Virtual teeth form, size, and setting will be done on the CAD software (Exocad Dental CAD 3.0, Exocad GmbH, Germany) according to jaw relation record.

The denture base extension and thickness will be designed on CAD software. The teeth will be exported in a separate file and the denture base will be exported in a separate stl file.

The virtual denture stl files will be sent to the 3D printer software (Chitubox software, CBD-Tech, china) where slicing of the file and adjustment of layers setting will be done.

The virtual denture will be sent to the 3D printer (photon 3d printer, ANYCUBIC 3D Printing, china) to be printed (printer has Y axis resolution: 1.25um and Layer resolution: 25 ~ 100um), Teeth will be printed alone using tooth-colored resin(dental sand, Harz labs, Russia) and base will be printed alone using pink resin(dental pink, HArzz lab, Russia), then it will be ethyl alcohol washed (99% ethyl alcohol) to remove excess resin. The teeth will be placed in their places in the denture base and secured using pink resin.

Post-curing for remaining uncured resin will be done using a post-curing chamber for 30 minutes (bre-lux power unit 2,bredent, united kingdom).

Regarding the maxillary denture:

Retention will be measured clinically by using a force gauge (weihang electronic gauge,weihang industries, china) for group A and group B at 0,1 and 3 months. A force gauge will be applied by fixing the chain at the center of the polished surface of the denture. The pull end of the force gauge will be connected to the denture to measure the retention. The force gauge will pull the denture vertically downward until denture retention will be lost, and the denture will move vertically. The force at which the denture dislodges will be recorded in grams. The pull-off procedure will be repeated 10 times to obtain 10 records for each elder, and then the mean of these records will be calculated.

Participants will answer a denture satisfaction questionnaire. Possible answers for each question and respective scores will be: unsatisfactory =0, regular =1, and good =2 (Rehmann et al., 2008) For group, A and group B denture base will be checked for accuracy of fit after scanning using a bench scanner with 1.3 megapixels dual camera and 10-micron accuracy (swing scanner, DOF inc, Korea) and will be compared to the virtual one planned on the master cast using metrology software (Geomagic Control X,3D systems, Canada). This will be done by the superimposition of the scanned printed or processed denture and the virtual reference denture. This will be done by selecting a point-to-point match and then the best fit function.

Color maps of the surface matching differences will be done. Areas that will be yellow to red in color will indicate impingement of the denture base with the cast. Areas that will be blue in color will indicate space between the denture base and cast. The ideal denture will show a color map that will be entirely green, giving a measurement value of 0, which will represent no processing deformation and an ideal adaptation of the denture base to the cast.

The results will be tabulated and statistically analyzed using SPSS Statistics Version 20 for Windows (SPSS, Inc., an IBM Company, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with good neuromuscular control and free of systemic diseases
* the edentulous ridge was covered with healthy firm and dense mucosa
* They have upper and lower edentulous healthy alveolar ridges with no remaining roots, no severe bony undercut, or local pathological lesions.
* patients had no previous dentures with a nearly equal edentulous period.

Exclusion Criteria:

* history of bad habits e.g. severe clenching.
* T.M.J disorders
* patients with xerostomia, high palatal vault, and short or hyperactive lips were excluded.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
accuracy of fit (adaptation) | 1 week
  the deviation of the denture fiitng surface from its corresponding cast will be measured using metrology software (GOM inspect,USA))
retention | 3 months
  retention will be measured using digital force gauge(weihang electronic gauge,weihang industries, china)
patient satisfaction | 3 months
  Participants will answer a denture satisfaction questionnaire. Possible answers for each question and respective scores will be: unsatisfactory =0, regular =1, and good =2 (Rehmann et al., 2008)

SECONDARY OUTCOMES:
retention over time period | 3 months
  change in denture retention over time period(0,1 and 3 months from denture insertion) will be measured for each group

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry,Suez Canal University, Bilbeis, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Goodacre BJ, Goodacre CJ, Baba NZ, Kattadiyil MT. Comparison of denture base adaptation between CAD-CAM and conventional fabrication techniques. J Prosthet Dent. 2016 Aug;116(2):249-56. doi: 10.1016/j.prosdent.2016.02.017. Epub 2016 Apr 23. PMID 27112416